CLINICAL TRIAL: NCT01126684
Title: EFFECTS OF ATORVASTATIN ON BLOOD PRESSURE AND URINARY ALBUMIN EXCRETION IN PATIENTS WITH ESSENTIAL HYPERTENSION
Brief Title: Effects of Atorvastatin on Blood Pressure and Urinary Albumin Excretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Lasaridis Anastasios, Professor of Internal Medicine and Nephrology, Aristotle University of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STAY
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-04

CONDITIONS: Hypertension; Hypercholesterolemia
Keywords: essential hypertension
MeSH Terms: conditions — Hypertension; Hypercholesterolemia; Essential Hypertension | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 10 mg of atorvastatin once daily for six months
  Arms: Atorvastatin
Drug: Placebo — placebo once daily for six months
  Arms: Placebo

SUMMARY:
To evaluate the possible effects of atorvastatin on ambulatory blood pressure, urinary albumin excretion, insulin resistance and arterial stiffness in hypertensive patients, beyond those on lipid profile. Glycemic parameters, "novel" cardiovascular risk factors and safety parameters will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C>130 or >160 mg/dL (depending on the total risk according to the most recent recommendations25).
* no previous hypolipidemic medication
* ability to provide Informed Consent.

Exclusion Criteria:

* pregnancy or lactation
* myocardial infarction or unstable angina within the past 6 months
* heart failure NYHA class III-IV
* renal disease (SCr>3 mg/dL or proteinuria>3g/d)
* liver disease
* history of malignancy
* history of drug or alcohol abuse
* treatment with corticosteroids
* any other condition with poor prognosis
* inability to provide Informed Consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure | Six months

SECONDARY OUTCOMES:
Urinary Albumin Excretion | Six months
Insulin Sensitivity | Six months
Arterial Stiffness | Six months
Urinary levels of nephrin | Six months
Urinary levels of podocalyxin | Six months
Urinary levels of Endothelin-1 | Six months
Urinary levels of Asymmetric Dimethylarginine | Six months
Urinary levels of indices of oxidative stress | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Lasaridis, MD, PhD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- AHEPA University Hospital of Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Kanaki AI, Sarafidis PA, Georgianos PI, Kanavos K, Tziolas IM, Zebekakis PE, Lasaridis AN. Effects of low-dose atorvastatin on arterial stiffness and central aortic pressure augmentation in patients with hypertension and hypercholesterolemia. Am J Hypertens. 2013 May;26(5):608-16. doi: 10.1093/ajh/hps098. Epub 2013 Feb 28. PMID 23449607